CLINICAL TRIAL: NCT00346099
Title: A Phase II Study to Determine the Efficacy and Safety of Panitumumab in Combination With Chemoradiotherapy for Unresectable or Locally Recurrent Adenocarcinoma of the Rectum With or Without Metastatic Disease
Brief Title: Study of Panitumumab Given First With Capecitabine and Oxaliplatin (CAPOX) and Then With Capecitabine and Radiation of the Pelvis for Treatment of Patients With Rectal Cancers That May or May Not Have Spread Beyond the Rectum
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Protocol closed based on new (and as yet unpublished) information from a phase II clinical trial.
Sponsor: NSABP Foundation Inc (Network)
Collaborators: Amgen (Industry)
Responsible Party: Norman Wolmark, MD, NSABP Foundation, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSABP FR-1
Record Dates: First submitted 2006-06-27; First posted 2006-06-29 (Estimated); Last update posted 2008-01-07 (Estimated); Status verified 2007-12

CONDITIONS: Rectal Cancer; Neoplasm Metastasis
Keywords: NSABP; panitumumab; rectal cancer; colorectal cancer; oxaliplatin; capecitabine; combined modality therapy; combined pelvic radiation therapy; Rectal cancer with or without metastasis
MeSH Terms: conditions — Rectal Neoplasms; Neoplasm Metastasis; Colorectal Neoplasms | interventions — Panitumumab; Capecitabine; Oxaliplatin; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Panitumumab with capecitabine and oxaliplatin (CAPOX) followed by
Drug: Panitumumab with capecitabine and radiation

SUMMARY:
Panitumumab is a monoclonal antibody. It works by attaching to a protein called epidermal growth factor receptor found on normal and cancer cells. When panitumumab attaches, it blocks another protein called epidermal growth factor (EGF) from attaching to the cell. This is important because, when EGF is blocked, a cell's growth slows down or stops. Panitumumab may also help radiation therapy work. Also because panitumumab is a fully-human antibody, it may be less toxic than other monoclonal antibodies made to block the EGF receptor. Chemotherapy, such as capecitabine and oxaliplatin, works to kill cancer cells directly. Capecitabine given during radiation helps radiation therapy work better. This study is being done to learn how rectal cancer tumors that are not removed surgically respond to treatment with panitumumab and chemotherapy given before radiation therapy begins followed by treatment with panitumumab and capecitabine given with radiation therapy.

DETAILED DESCRIPTION:
Colorectal cancers express EGF and/or EGFR mRNA in 66% of primary tumors, 44% of adjacent mucosa, and up to 62% of positive lymph nodes. Patients enrolled in NSABP FR-1 will begin therapy with the anti-EGFR antibody panitumumab--which has shown single-agent activity in colorectal cancer patients--in combination with CAPOX, an effective treatment for patients with advanced colorectal cancer, with the convenience of using an oral fluoropyrimidine (capecitabine.) The intent with this first phase is to expose distant metastases to the agents early and to shrink the tumor before giving radiation therapy. After chemotherapy, radiotherapy with capecitabine and panitumumab will be given to destroy the primary tumor. Panitumumab is added to the radiochemotherapy regimen because data showed positive results when another anti-EGFR antibody was added to radiotherapy in patients with head and neck cancer. This approach aims to improve neoadjuvant combined modality therapy for rectal cancer; it should provide effective therapy for eligible patients and valuable information about clinical tumor response rates and treatment tolerability, which, if favorable, may be used to develop future Phase III trials.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic diagnosis of rectal cancer (adenocarcinoma)
* Must have rectal cancer that is:

  * locally advanced and considered not to be curable by surgery
  * recurrent (if it was treated before by surgical removal of the tumor)
  * present along with small-volume metastasis
* Evidence of adequate organ function (such as liver, kidneys, etc.)
* Must be able to swallow tablets
* Able to perform an adequate level of physical activity

Exclusion Criteria:

* Diagnosis of rectal cancer other than adenocarcinoma
* Patients who are candidates for surgical removal of metastatic and/or locally advanced disease
* Patients who have received previous treatments for the current cancer
* Chronic liver disease or recurrent viral hepatitis
* Any previous pelvic radiation therapy and/or any previous chemotherapy with oxaliplatin or epidermal growth factor receptor inhibitors
* Central nervous system metastases
* Active inflammatory bowel disease
* Current clinically significant abnormal peripheral nerve disease
* Active heart disease, including blocked blood vessels, recent heart attack, history of congestive heart failure, or abnormal heart beat
* Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-06; Study Completion 2007-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with clinical complete response rate in tumor in the pelvis at 4 to 6 weeks after completion of radiation therapy

SECONDARY OUTCOMES:
Percentage of patients with pathologic complete response rate of the primary rectal tumor and resected regional lymph nodes(tissue removed at the time of surgery)
Percentage of patients whose surgical evaluation following therapy indicates candidacy for resection
Percentage of patients who have progressive disease in the pelvis from the time of study entry to 2 years
The toxicity of panitumumab in combination with chemotherapy and in combination with chemoradiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — National Surgical Adjuvant Breast and Bowel Project Foundation, Inc.